CLINICAL TRIAL: NCT07304349
Title: Prospective Multicenter Field Study for Rapid Diagnostic Tests Evaluation for Timely Detection of Chronic Chagas Disease in Public Health Sites in Argentina.
Brief Title: Prospective Evaluation of Rapid Diagnostic Tests for Trypanosoma Cruzi Infection
Status: Recruiting | Type: Observational
Sponsor: Instituto Nacional de Parasitologia Dr. Mario Fatala Chaben (Other Government)
Collaborators: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Sponsor
Other Study IDs: CH-RDT-009
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Chagas
Keywords: serological diagnosis; diagnostic performance; immunochromatography; neglected tropical diseases
MeSH Terms: conditions — Neglected Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Up to 50 µl capillary blood or ≥1 ml venous blood (EDTA) for RDTs. 3-8 ml venous blood (serum) for reference tests.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chagas disease (CD) is the most significant endemic zoonosis in Argentina. Two-thirds of affected individuals live in urban areas but only 10% globally are aware of their infection. Diagnosing Chronic Chagas (CCD) requires at least two serological tests, often limited to reference laboratories, creating logistical and economic challenges that delay timely diagnosis and treatment. Although primary health care (PHC) could address most health needs, the availability of Rapid Diagnostic Tests (RDTs) for CCD is limited in endemic countries due to regulatory and commercial barriers. In 2023, in a laboratory evaluation (Instituto Nacional de Parasitología, INP-ANLIS) we demonstrated that performance of six commercial RDTs available in Argentina were similar to reference methods, suggesting their potential for CCD diagnosis use (standard diagnostic", PAHO, 2018). Evaluation of RDTs in field studies across different clinical and epidemiological contexts is mandatory to provide recommendations for their use in CCD diagnosis. In this sense, independent prospective studies should be conducted to evaluate RDTs tests performances using direct blood samples under field conditions in different health care facilities and epidemiological scenarios. Moreover, trials conducted in different countries should be comparable with each other, so this protocol, produced according to STARD 2015 standards, is proposed as a complement to the PAHO (2025) recommendations. These RDT evaluation studies have the ultimate objective of incorporating them into diagnostic algorithms for better access to treatment and care strategy for patients with chronic CD.

DETAILED DESCRIPTION:
Background and Rationale: Chagas disease (CD) is the most important endemic zoonosis in Argentina. Most affected individuals live in urban areas, and only a minority are aware of their diagnosis. Current diagnostic methods require multiple serological tests, often available only at reference laboratories, causing delays in access to diagnosis and treatment. Rapid diagnostic tests (RDTs) offer a potential solution for timely detection in primary health care settings, but field validation studies are needed.

Hypothesis: RDTs evaluated will detect infection with sensitivity >90% and specificity >95%.

Primary Objectives:

To evaluate the performance of two RDTs for supporting the management of chronic T. cruzi infection.

To identify a high-performance diagnostic algorithm incorporating RDTs at the point of care (POC).

Secondary Objectives Assess concordance of RDTs across sample types (capillary, venous, serum). Assess concordance between RDTs and the current diagnostic algorithm. Evaluate usability of RDTs for CD.: Estimate cost-effectiveness of implementing RDT-based algorithms in Argentina.

Assess whether RDTs improve access to diagnosis. Estimate prevalence of T. cruzi infection in the study population. Primary Endpoints Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) of RDTs compared to the standard reference algorithm.

Diagnostic accuracy of RDT-based algorithms (Youden's index). Secondary Endpoints Concordance between sample types and between RDTs and reference algorithm (Cohen's Kappa).

Usability scores of RDTs. Incremental cost-effectiveness ratio (ICER) of RDT-inclusive algorithms. Accessibility scores (socioeconomic profile, costs, transport time, food, income loss).

Proportion of positive samples among total analyzed. Study Design: Prospective, multicenter, observational, cross-sectional field study.

Study Sites: Hospitals Mercante, Paroissien, Gutiérrez, and other health centers in Buenos Aires Province.

Study Population: Inclusion: Pregnant women, blood donors, transplant recipients, suspected chronic T. cruzi infection, >10 months of age, with informed consent/assent.

Exclusion: Previous antiparasitic treatment, immunocompromised individuals, or conditions preventing protocol implementation/interpretation.

Samples: Up to 50 µl capillary blood or ≥1 ml venous blood (EDTA) for RDTs. 3-8 ml venous blood (serum) for reference tests. Sample Size: Estimated N = 3,234, including 152 positive samples. Index Tests: Two Commercially available RDTs selected based on availability, cost, and performance. Conducted at POC per manufacturer's instructions. Results used exclusively for research.

Reference Standard: Infection: reactive results from two distinct serological tests (ELISA, HAI, IFA).

Non-infection: non-reactive results from two tests. Laboratory results will be blinded to RDT results and will serve as the patient care standard.

Data Collection: Clinical and epidemiological data collected. RDT results recorded at POC; reference test results recorded at site laboratories.

Duration 24 months. Ethics: Approved by the INP ANLIS Ethics Committee and the Central Ethics Committee of the Ministry of Health of the Province of Buenos Aires.

Funding: Approved by hospital directors in the province of Buenos Aires. Funded by the National University of José C. Paz (UNPAZ) and the National University of La Matanza (UNLaM). Approved by the Directorate of Epidemiological Surveillance and Outbreak Control. Chagas Prevention and Control Programme. Ministry of Health of the Province of Buenos Aires. (Provincial Programme against Chagas). Funded by FIND, Foundation for Innovative New Diagnostics, Geneva, Switzerland.

ELIGIBILITY:
Inclusion Criteria: Pregnant women, blood donors, transplant recipients, suspected chronic T. cruzi infection, >10 months of age, with informed consent/assent.

Exclusion Criteria: Previous antiparasitic treatment, immunocompromised individuals, or conditions preventing protocol implementation/interpretation.

Min Age: 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited within the framework of healthcare provision. Participation in the study will be offered to individuals over 10 months of age, or their parents or guardians where applicable, who attend study centres or participate in health promotion activities or territorial testing initiatives organised by INP ANLIS, the Ministry of Health of the Province of Buenos Aires, UNPAZ or UNLaM.
Sampling Method: Non-Probability Sample
Enrollment: 3234 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the performance of two rapid diagnostic tests (RDTs) to support the treatment of chronic T. cruzi infection. Identify a high-performance diagnostic algorithm that incorporates point-of-care (POC) RDTs. | From August 2025 to May 2027.
  Point estimates (with 95% CI) of sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of two commercially available T. cruzi RDTs, using the current EC diagnostic algorithm as the reference method.
  These measures are proportions expressed on a scale ranging from 0 to 1, where higher values indicate better diagnostic performance.
  To evaluate the overall diagnostic performance of the RDT-based algorithm, Youden's Index (unabbreviated: Youden's Index) will be calculated. Youden's Index is defined as sensitivity + specificity - 1 and is measured on a scale ranging from -1 to +1, where higher values indicate better discriminatory ability.

SECONDARY OUTCOMES:
Estimate the concordance of RDTs for T. cruzi using different types of samples. | From August 2025 to April 2027
  Agreement between RDTs for T. cruzi results obtained from capillary, venous, and serum blood samples will be evaluated using Cohen's Kappa coefficient. Cohen's Kappa is measured on a scale ranging from -1 to +1, where higher values indicate stronger agreement beyond chance, with +1 indicating perfect agreement, 0 indicating agreement equivalent to chance, and negative values indicating agreement worse than chance.
Estimate the concordance between the RDTs for T. cruzi and the current diagnostic algorithm for CD. | from August 2025 to June 2027
  Agreement between T. cruzi RDTs and the current diagnostic algorithm for CD will also be assessed using Cohen's Kappa coefficient. The scale ranges from -1 to +1, and higher values represent better concordance between diagnostic approaches.
Evaluate the usability of T. cruzi RDTs. | August 2025 to August 2027
  Usability of the RDTs will be evaluated using the System Usability Scale (SUS) developed by FIND specifically for the evaluation of RDTs for T. cruzi. The SUS is measured on a scale ranging from 4 (minimum) to 10 (maximum), where higher scores indicate better usability and a more favorable user experience.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita M. C. Bisio, PhD, Study Chair — National Council of Scientific and Technical Research, Argentina
Locations (4):
- Argentina (4):
  - Hospital Mercante, Buenos Aires, Buenos Aires
  - Hospital Gutierrez, Buenos Aires, Buenos Aires
  - Hospital Paroissien, Isidro Casanova, Buenos Aires
  - Dispositivos Territoriales, Olmos, La Plata, Buenos Aires

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol